CLINICAL TRIAL: NCT01926444
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase 2a Proof-of-Concept Study of GIC-1001 for the Management of Visceral Pain in Subjects Undergoing Sedation-Free, Full Colonoscopy
Brief Title: A Phase 2a, Proof-of-Concept Study of GIC-1001 in the Management of Visceral Pain During Sedation-Free, Full Colonoscopy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: gicare Pharma Inc. (Industry)
Collaborators: JSS Medical Research Inc. (Industry); Algorithme Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: GIC13-01
Record Dates: First submitted 2013-08-08; First posted 2013-08-21 (Estimated); Results first posted 2019-05-08 (Actual); Last update posted 2019-05-08 (Actual); Status verified 2019-05

CONDITIONS: Pain; Cancer; Colonic Diseases
Keywords: colonoscopy; sedation-free; colorectal cancer; CRC screening; prevention; analgesia; colonic; kappa; opioid agonist; pain management; oral; hydrogen sulfide; peripheral
MeSH Terms: conditions — Pain; Neoplasms; Colonic Diseases; Colorectal Neoplasms; Agnosia | interventions — trimebutine 3-thiocarbamoylbenzenesulfonate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- GIC-1001 low dose (Experimental): GIC-1001 , 250 mg TID during 3 consecutive days + a last, 10th dose in the morning of Day 4 (colonoscopy day)
  Interventions: Drug: GIC-1001
- GIC-1001 mid-dose (Experimental): GIC-1001 , 375 mg TID during 3 consecutive days + a 10th dose in the morning of day 4 (colonoscopy day)
  Interventions: Drug: GIC-1001
- GIC-1001 , high dose (Experimental): GIC-1001 , 500 mg TID during 3 consecutive days + a 10th dose in the morning of day 4 (colonoscopy day)
  Interventions: Drug: GIC-1001
- GIC-1001 matching placebo (Placebo Comparator): Placebo, TID during 3 consecutive days, + a 10 th dose in the morning of day 4 (colonoscopy day)
  Interventions: Drug: GIC-1001

INTERVENTIONS:
Drug: GIC-1001 — GIC-1001 oral tablet, white-coated, to be taken with water
  Other Names: trimebutine 3-thiocarbamoylbenzenesulfonate; TB-905-02

SUMMARY:
GIC-1001 is a novel, orally-administered, colonic analgesic drug developed as an alternative to i.v. sedation during full colonoscopy. It will be evaluated for efficacy and safety in a multi-center, randomized, double-blind, placebo controlled, dose-ranging, proof of concept Phase 2a trial. Up to 240 patients will receive one of 3 doses of GIC-1001 or its matching placebo. A pharmacokinetic evaluation will be carried out on a subset of patients (N: 24).

DETAILED DESCRIPTION:
1. Study Objectives

   1.1 Primary objective: The primary objective of this Phase IIa study is to establish clinical Proof-of-Concept (POC) by providing clinically and statistically significant evidence that GIC-1001 is safe and effective in managing visceral pain in male and female patients who undergo sedation-free, full colonoscopy for preventive purposes.

   1.2 Secondary objectives: Secondary objectives will include the selection of the optimal dose of GIC-1001 from a safety/efficacy ratio point of view, establish a preliminary safety profile of the drug in patients, and obtain a preliminary general efficacy profile of GIC-1001 by assessing various secondary endpoints
2. Study Endpoints

   2.1 Primary endpoints:

   Visceral pain will be assessed using a 100-mm VAS, measured at various times and anatomical segments (N: 8) throughout the colon, i.e.:
   1. Prior to intra-rectal insertion of the endoscope;
   2. After insertion through the anus;
   3. After passage through the rectosigmoid segment;
   4. Immediately after passage through the splenic flexure;
   5. Immediately after passage through the hepatic flexure;
   6. Once the caecum is reached;
   7. Immediately after passage through the splenic flexure during scope withdrawal; and
   8. At the end of the procedure, once the colonoscope has been completely removed. Any additional episodes of pain experienced by the patient will also be assessed using the 100-mm VAS scale.

   The area under the curve (AUC) calculated from all serial measurements made will be used for statistical purposes, where the length of inserted colonoscope determines the VAS measurement's location.

   2.2 Secondary endpoints:
   1. Overall pain perception (100-mm VAS) at the end of the procedure;
   2. Time to reach the caecum with the endoscope (intubation time from rectum to caecum defined as time-to-caecum);
   3. Total examination time, defined at the time from introduction to removal of the colonoscope;
   4. Percentage of completed procedures;
   5. Endoscopist's perception of the adequacy of analgesia, difficulty of insertion, and amount of colonic spasm on insertion and withdrawal (five-point Likert scale);
   6. Use of rescue sedation (i.e. midazolam or midazolam followed by fentanyl)
   7. Safety as assessed by the incidence of treatment emergent adverse effects during the procedure and for 30 days after;
   8. Plasma determination of trimebutine and N-desmethyl-trimebutine moieties at GIC-1001 plasmatic steady state;
   9. Patient satisfaction with treatment (five-point Likert scale);
   10. Patient' willingness for repeat colonoscopy in the future (five-point Likert scale); and
   11. Safety of GIC-1001.
3. Study Design This is a randomized, double-blind, placebo-controlled parallel design 4-treatment arms study. Eligible patients will be randomized in a 1:1:1:2 ratio to one of 4 treatment arms: low (250 mg), mid (375 mg) or high (500 mg) dose of GIC-1001, or matching placebo. All potential study subjects will be screened and assessed for eligibility within maximum two (2) weeks prior to randomization. Bowel preparation will be performed using a polyethylene glycol (PEG) based regimen the night before the actual procedure.
4. Number of Clinical Sites: This trial will be conducted in both Canada and USA. Up to ten (10) clinical sites will participate in this trial. The lead Investigator for this trial is Dr Mark V. Larson MD, Head of Digestive Endoscopy, Mayo Clinic, Rochester MN, USA
5. Study population and sample size: Approximately 240 patients will be randomized in this study. Male and female patients having an indication for full colonoscopy, mainly for colorectal cancer screening and surveillance. Only naïve subjects, i.e. who never underwent colonoscopy before, will be eligible.
6. Inclusion Criteria See Eligibility Section
7. Exclusion Criteria See Eligibility Section
8. Study Drugs Administration and Schedule:

   GIC-1001, or its matching placebo will be administered as follows:
   1. One tablet TID on an empty stomach for three (3) consecutive days prior to colonoscopy.
   2. Last dose taken at the clinical site at least one (1) hour prior to beginning of procedure (endoscope insertion).
   3. Bowel preparation to be performed using PEG based regimen the day before the actual procedure.
   4. Three (3) different GIC-1001 dose levels will be studied:

      * 250 mg TID
      * 375 mg TID
      * 500 mg TID
      * Matching placebo TID
9. Concomitant Medications

   9.1 Prior to colonoscopy, the following medication will be permitted: Aspirin (ASA) at low levels for cardiovascular health, if dose and regimen stable for the last 6 months prior to colonoscopy.

   9.2 The following medications and foods will be prohibited:
   * Any prescription chronic analgesic narcotic, anti-spasmodic, anti-inflammatory medications are forbidden for 30 days prior to screening. (i.e. Washout ≥ 30 days)
   * Selective Serotonin Re-uptake Inhibitors (SSRIs) are forbidden for 30 days prior to screening, unless patient has been on a stable dose for 3 consecutive months prior to screening.
   * Over-the-counter analgesics, or anti-inflammatory medication, oral or topical used for acute pain treatment must be washed out for ≥ 7days prior to screening.
   * Acute or as needed prescription or non-prescription anti-inflammatory and/or analgesic treatment within one (1) week prior to colonoscopy.
   * Use of bowel stimulant laxatives, such bisacodyl, within one (1) week preceding randomization.
   * Use of antidiarrheic medication, such as diphenoxylate, loperamide, kaopectate or bismuth salts, within one (1) week preceding randomization.
   * Administration of barium enema within two (2) weeks preceding randomization.
   * Colonic irritant beverages or foods, such as caffeine-containing beverages (e.g. coffee, Coca-Cola), spices, as well as foods containing seeds (i.e. tomatoes, strawberries, kiwis, raspberries) within 24 hours preceding colonoscopy.
   * Use of any other investigational drug is prohibited unless discontinued, within at least 30 days prior to randomization.
   * Additionally, Prior and Concomitant Medications are to be recorded in the CRF starting 30 days prior to Screening Visit CLV1.
10. Efficacy Evaluation: Colonic analgesic clinical efficacy of GIC-1001 will be measured using a continuous, horizontal 100-mm VAS, at pre-determined times and colonic anatomical segments. At least 8 measurements will be done by the participating patients themselves (see Primary Endpoint section). Subjects will receive proper instructions on the use of the VAS prior to colonoscopy. Overall experience of visceral pain (if any) will be evaluated using the AUC constructed from all calculated VAS self-measurements for each patient. Additional, secondary, efficacy endpoints will also be measured, including time-to-caecum, colonoscopy completion rate and antispasmodic activity.
11. Safety Evaluation: Safety will be assessed using the performance of physical exams, ECG, various laboratory safety tests and the occurrence of adverse events. AEs will be mapped to MedDRA, version 16.
12. Sample Size Considerations: It has been reported in the medical literature that a MCID range of 10-15 mm on the 100-mm VAS is clinical significant in the evaluation of colonoscopy-related visceral pain. Using this value, with an alpha of 0.05 and a beta of 0.9, about 50 patients would be needed in each active arm considering a 90-patient placebo arm. Total study sample size is then estimated at approximately 240 randomized patients.
13. Statistical Analysis: The primary outcome measure will be the mean 100-mm VAS AUC in each treatment arm.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated written Informed Consent obtained.
2. Males or females.
3. Aged 40-75 years.
4. Indication for full colonoscopy for colorectal cancer screening or investigation, including subjects presenting suggestive symptoms and who need a differential diagnosis.
5. Colonoscopy naïve subjects, i.e. who never underwent colonoscopy before, will be eligible, as well as non-naïve subjects who have previously undergone unsedated colonoscopy , or who had sedated colonoscopy at least 10 years prior (i.e. ≥ 10 years) to enrolment
6. Eligible for a procedure without sedation.
7. Able to complete questionnaires and use a Visual Analog Scale (VAS), including sufficient English, French or Spanish speaking skills as well as adequate eyesight and hearing
8. BMI ≥ 19, BMI ≤ 40 kg/m2.

Exclusion Criteria:

1. Known allergy or intolerance to trimebutine (Modulon® or generic).
2. Known allergy or intolerance to sulfur-containing drugs (e.g. N-acetylcysteine or captopril).
3. Previous gastrointestinal or gynecologic surgery, e.g. ileostomy, pelvic surgery,; however, patients with an appendectomy are eligible.Patients who have had a tubal ligation at least 10 years prior (i.e. ≥ 10 years) to enrolment are also eligible.
4. Diagnosed Inflammatory Bowel Disease (IBD).
5. Visceral hypersensitivity conditions such as Irritable Bowel Syndrome (IBS).
6. Clinically significant renal and/or hepatic impairment.
7. History of peritonitis.
8. Known severe diverticular disease.
9. Severe diverticulosis as documented by prior imaging series
10. Known or suspected stenosis of the colon.
11. Chronic pain syndrome such as fibromyalgia and endometriosis.
12. Any clinically-relevant abnormality identified on the screening, history, physical examination, 12-lead ECG or laboratory examination, which would, in the Investigator's opinion, preclude the administration of investigational drug product, GIC1001
13. Unexpected and significant visceral pain reported by subject prior to colonoscopy.
14. Dementia.
15. Diagnosed clinically significant psychiatric illness, including severe anxiety disorders that may affect the subject's perception of visceral pain or ability to participate in the study.
16. Patient is a lactating female.
17. Female is of childbearing potential sexually active who are unwilling or unable to use an acceptable method of contraception (which includes oral or implanted contraceptives, IUD, female condom, diaphragm with spermicide, cervical cap, use of a condom by the sexual partner or sterile sexual partner) throughout the duration of the study and 1 month following study completion.
18. Female is of childbearing potential, sexually abstinent who does not agree to continue abstinence or to use one of the acceptable methods of birth control should sexual activity commence.
19. Any serious medical condition that could increase the risk of adverse reactions with trimebutine.
20. Participation in another experimental drug trial within 30 days of randomization.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 308 (Actual)
Dates: Start 2013-07; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark V Larson, MD, Study Chair — Mayo Clinic, Rochester, MN, USA; Michael DeMicco, MD, Principal Investigator — Anaheim Clinical Trials, Anaheim, CA, USA; Mark Lamet, MD, Principal Investigator — The Center of GI Disorders, Hollwood, FL, USA; Taddese Desta, MD, Principal Investigator — Precision Research Institute, San Diego, CA, USA; Cynthia Schaeffer, MD, Principal Investigator — Precision Research Institute, Chula Vista, CA, USA; Vivek Gumaste, MD, Principal Investigator — Montefiore Medical Center, NY, USA; Theadore Ptak, MD, Principal Investigator — Toronto Digestive Disease Associates, Toronto, ON, Canada; Anand Sahai, MD, Principal Investigator — Clinique 1037, Montreal, QC, Canada; Umedchandra Shah, MD, Principal Investigator — Mid-Atlantic Medical Research Centers, Hollyword, MD, USA; Suryakanth R. Gurudu, MD, Principal Investigator — Mayo Clinical, Scottsdale Arizona; Robert Enns, MD, Principal Investigator — GIRI (GI Research Institute), Vancouver, Canada; Narayanachar S Murali, MD, Principal Investigator — Gastroenterology Associates of Orangeburg, SC, USA; Vishal Gupta, MD, Principal Investigator — Avail Clinical Research LLC; Albert Cohen, MD, Principal Investigator — Spécialistes MD Specialists; Vitaly Fishbein, MD, Principal Investigator — PharmaTrials; Dennis Riff, MD, Study Director — Anaheim Clinical Trials
Locations (15):
- United States (11):
  - Mayo Clinic, Scottsdale, Arizona
  - Anaheim Clinical Trials, Anaheim, California
  - Precision Research Institute, Chula Vista, California
  - Precision Research Institute, San Diego, California
  - Avail Clinical Research LLC, DeLand, Florida
  - The Center for GI Disorders, Hollywood, Florida
  - Mid-Atlantic Medical Research Centers, Hollywood, Maryland
  - Mayo Clinic Rochester, Rochester, Minnesota
  - PharmaTrials, Hillsborough, New Jersey
  - Montefiore Medical Center, The Bronx, New York
  - Gastroenterology Associates of Orangeburg, Orangeburg, South Carolina
- Canada (4):
  - GIRI (GI Research Institute), Vancouver, British Columbia
  - Toronto Digestive Disease Associates, Toronto, Ontario
  - Clinique 1037, Montreal, Quebec
  - Spécialistes MD Specialists, Montreal, Quebec

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient enrolled: 25 JULY 2013; Last patient completed: 03 MARCH 2014
Pre-assignment Details: A total of N=37 subjects were screen failures and were not randomized (total randomized = 271/308). Of those randomized, N=268 subjects received at least one dose of study drug, and were included in the Safety Population.
Period: Overall Study
Arm/Group | GIC-1001 Low Dose | GIC-1001 Mid-dose | GIC-1001 , High Dose | GIC-1001 Matching Placebo
Started | 56 | 52 | 57 | 103
Completed | 56 | 52 | 53 | 101
Not Completed | 0 | 0 | 4 | 2
Not completed — Colonoscopy not performed | 0 | 0 | 4 | 2

BASELINE CHARACTERISTICS:
Population: Demographics provided for the Full Analysis Set (FAS; N=262), defined as all randomized patients who received at least one dose of study drug, had a baseline and at least one post-baseline VAS rating.
Groups:
- Total: Total of all reporting groups
Arm/Group | GIC-1001 Low Dose | GIC-1001 Mid-dose | GIC-1001 , High Dose | GIC-1001 Matching Placebo | Total
Number analyzed (Participants) | 56 | 52 | 53 | 101 | 262
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.35 (7.04) | 54.68 (5.81) | 53.74 (6.89) | 54.32 (7.32) | 54.28 (6.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 19 | 19 | 35 | 89
  Male | 40 | 33 | 34 | 66 | 173
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian/Oriental | 6 | 1 | 5 | 5 | 17
  Black | 10 | 10 | 8 | 23 | 51
  Caucasian | 31 | 28 | 30 | 51 | 140
  Hispanic | 9 | 13 | 9 | 20 | 51
  Other | 0 | 0 | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Measurements of Visceral Pain, Using a 100-mm Visual Analog Scale (VAS)
Description: The Primary Outcomes Measure was the pain VAS 100-mm AUC (0mm = no pain; 100mm = worst pain), constructed from serial pain VAS measurements performed during colonoscopy. At least 8 pain VAS measurements were made, and the length of the colonoscope inserted (or removed on the way out) was recorded at every measurement. The X-axis of the VAS versus anatomical locations was defined accordingly: each VAS value corresponded to a relative length of inserted colonoscope (d/2Lc) of the X axis, where d was the actual length of the inserted colonoscope and 2Lc represented twice the total length of the colon examined (Lc). Before scope insertion the X value equaled zero. Once the caecum was reached, the X value was 0.5. Upon complete removal of the endoscope, the X value was 1. This allowed standardization of colonic length between study subjects. Visceral pain AUC (mm) was calculated from all serial measurements, where the length of inserted colonoscope determined the VAS measurement's location
Time Frame: Assessed at different anatomical locations: (1) before colonoscopy, (2) insertion of scope in anus, (3) at rectosigmoid flexure, (4) at splenic flexure, (5) at hepatic flexure, (6) at caecum, (7) at splenic flexure on way back, (8) after colonoscopy.
Population: Primary endpoint assessed in the FAS (randomized patients who received at least one dose of study drug, had a baseline and at least one post-baseline VAS rating; N=262) and PP analysis sets (randomized patients in the FA population with ≥80% treatment compliance, who had at least 6/8 VAS ratings and no major protocol deviations; N=213)
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | GIC-1001 Low Dose | GIC-1001 Mid-dose | GIC-1001 , High Dose | GIC-1001 Matching Placebo
Number analyzed (Participants) | 56 | 52 | 53 | 101
mm
  AUC- censorsed (standardized); FAS | 22.27 (16.31) | 18.93 (13.11) | 23.31 (16.12) | 22.22 (16.44)
  AUC LOCF (standardized); FAS | 25.5 (19.77) | 23.44 (18.7) | 27.73 (18.00) | 27.55 (20.00)
  AUC- censorsed (standardized); PP: number analyzed (Participants) | 48 | 43 | 42 | 80
  AUC- censorsed (standardized); PP | 20.79 (16.56) | 17.6 (13.31) | 24.61 (17.18) | 22.03 (16.35)
  AUC LOCF (standardized); PP: number analyzed (Participants) | 48 | 43 | 42 | 80
  AUC LOCF (standardized); PP | 20.96 (16.41) | 17.63 (13.29) | 24.8 (17.17) | 22.00 (16.28)
Statistical Analysis 1: Comparison: GIC-1001 Low Dose vs GIC-1001 Mid-dose vs GIC-1001 , High Dose vs GIC-1001 Matching Placebo; AUC- censorsed (standardized); FAS; Test type: Other; p = 0.506, ANOVA
Statistical Analysis 2: Comparison: GIC-1001 Low Dose vs GIC-1001 Mid-dose vs GIC-1001 , High Dose vs GIC-1001 Matching Placebo; AUC LOCF (standardized); FAS; Test type: Other; p = 0.299, ANOVA
Statistical Analysis 3: Comparison: GIC-1001 Low Dose vs GIC-1001 Mid-dose vs GIC-1001 , High Dose vs GIC-1001 Matching Placebo; AUC Censored (Standardized)- PP Population; Test type: Other; p = 0.234, ANOVA
Statistical Analysis 4: Comparison: GIC-1001 Low Dose vs GIC-1001 Mid-dose vs GIC-1001 , High Dose vs GIC-1001 Matching Placebo; AUC LOCF (Standardized)- PP Population; Test type: Other; p = 0.219, ANOVA

2. Secondary Outcome: Time to Caecum
Description: Time to Caecum is the time taken by the physician to reach the caecum with the colonoscope, from the insertion in the anus. Time to Caecum was measured during colonoscopy, for which total duration of colonoscopy ranged between a minimum of 5.00 and a maximum of 50.10 minutes.
Time Frame: From the time of introduction of the colonoscope, to removal of colonoscope. Range of duration of colonoscopy 5.00- 50.10 minutes.
Population: FAS (randomized patients who received at least one dose of study drug, had a baseline and at least one post-baseline VAS rating; N=262)
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | GIC-1001 Low Dose | GIC-1001 Mid-dose | GIC-1001 , High Dose | GIC-1001 Matching Placebo
Number analyzed (Participants) | 56 | 52 | 53 | 101
minutes | 8.47 (4.75) | 6.51 (2.67) | 9.22 (6.10) | 8.04 (5.33)
Statistical Analysis 1: Comparison: GIC-1001 Low Dose vs GIC-1001 Mid-dose vs GIC-1001 , High Dose vs GIC-1001 Matching Placebo; Time to Caecum; Test type: Other; p = 0.047, Chi-squared

3. Secondary Outcome: Colonoscopy Completion Rate (%)
Description: Qualitative outcome: colonoscopy completion is defined as a procedure performed entirely, from initial anal insertion, reaching of caecum, and complete removal of the scope. Completion rate is then the number of patient (%) with a complete colonoscopy (up to the caecum) divided by the number of trial participants.
Time Frame: Number of patients during trial with a complete colonoscopy, where the scope has reached the caecum during the colonoscopy. Range of duration of colonoscopy 5.00- 50.10 minutes.
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | GIC-1001 Low Dose | GIC-1001 Mid-dose | GIC-1001 , High Dose | GIC-1001 Matching Placebo
Number analyzed (Participants) | 56 | 52 | 53 | 101
Participants | 56 | 52 | 51 | 101
Statistical Analysis 1: Comparison: GIC-1001 Low Dose vs GIC-1001 Mid-dose vs GIC-1001 , High Dose vs GIC-1001 Matching Placebo; Test type: Other; p = 0.047, Chi-squared

4. Secondary Outcome: Safety-Plasma Concentrations of Trimebutine and N-Desmethyl-Trimebutine
Description: A pharmacokinetic (PK) analysis was carried out on the first 24 patients randomized, equally distributed between treatment groups; 18 patients were assigned to active treatment
Time Frame: Day 4 prior to colonoscopy.
Population: Trimebutine and N-Desmethyl-Trimebutine plasma concentrations were assessed in all arms, with the exception of placebo
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | GIC-1001 Low Dose | GIC-1001 Mid-dose | GIC-1001 , High Dose | GIC-1001 Matching Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 0
ng/mL
  Plasma Concentration- Trimebutine | 5.17 (1.96) | 8.80 (3.55) | 16.22 (7.32) |
  Plasma Concentration-N-Desmethyl-Trimebutine | 174.5 (130.1) | 440.98 (546.53) | 389.18 (166.42) |

5. Secondary Outcome: Total Examination Time (Colonoscopy)
Description: Defined as the time from endoscope insertion to complete removal of the endoscope; measured in minutes
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | GIC-1001 Low Dose | GIC-1001 Mid-dose | GIC-1001 , High Dose | GIC-1001 Matching Placebo
Number analyzed (Participants) | 56 | 52 | 53 | 101
minutes | 15.82 (7.06) | 13.05 (6.22) | 15.52 (8.08) | 14.61 (7.58)

6. Secondary Outcome: Endoscopist's Perception of Colonoscopy- Adequacy of Analgesia, Difficulty of Insertion and Withdrawal
Description: Endoscopist's perception of the adequacy of analgesia, difficulty of insertion and withdrawal measured on a five-point Likert scale: Strongly Agree, Agree, Agree nor Disagree, Disagree, Strongly Disagree
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | GIC-1001 Low Dose | GIC-1001 Mid-dose | GIC-1001 , High Dose | GIC-1001 Matching Placebo
Number analyzed (Participants) | 56 | 52 | 53 | 101
Participants
  Adequate Analgesia: Strongly Agree | 20 | 18 | 16 | 33
  Adequate Analgesia: Agree | 14 | 21 | 17 | 30
  Adequate Analgesia: Agree nor Disagree | 8 | 3 | 4 | 10
  Adequate Analgesia: Disagree | 9 | 6 | 11 | 16
  Adequate Analgesia: Strongly Disagree | 5 | 4 | 5 | 12
  Difficult Insertion: Strongly Agree | 3 | 2 | 3 | 5
  Difficult Insertion: Agree | 7 | 6 | 7 | 24
  Difficult Insertion: Agree nor Disagree | 6 | 5 | 4 | 10
  Difficult Insertion: Disagree | 22 | 19 | 21 | 31
  Difficult Insertion: Strongly Disagree | 18 | 20 | 18 | 31
  Difficult Withdrawal: Strongly Agree | 0 | 0 | 0 | 1
  Difficult Withdrawal: Agree | 0 | 1 | 2 | 2
  Difficult Withdrawal: Agree nor Disagree | 0 | 1 | 0 | 1
  Difficult Withdrawal: Disagree | 19 | 18 | 15 | 29
  Difficult Withdrawal: Strongly Disagree | 37 | 32 | 36 | 68

7. Secondary Outcome: Endoscopist's Perception of Colonoscopy- Amount of Colonic Spasm on Insertion and Withdrawal
Description: Endoscopist's perception of the amount of colonic spasm on insertion and withdrawal measured on five-point Likert scale according to the following: Strongly Agree, Agree, Agree nor Disagree, Disagree, Strongly Disagree
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | GIC-1001 Low Dose | GIC-1001 Mid-dose | GIC-1001 , High Dose | GIC-1001 Matching Placebo
Number analyzed (Participants) | 56 | 52 | 53 | 101
Participants
  Colonic Spasm insertion: Absent | 33 | 33 | 33 | 59
  Colonic Spasm insertion: Present and minimal # (1 spasm) | 11 | 7 | 11 | 20
  Colonic Spasm insertion: Present and moderate #(2-3 spasms) | 8 | 10 | 6 | 11
  Colonic Spasm insertion: Present and high # (4-5 spasms) | 2 | 2 | 1 | 9
  Colonic Spasm insertion: Present and very high (>5 spasms) | 2 | 0 | 2 | 2
  Colonic Spasm WIthdrawal: Absent | 41 | 40 | 45 | 83
  Colonic Spasm WIthdrawal: Present and minimal # (1 spasm) | 11 | 8 | 6 | 14
  Colonic Spasm WIthdrawal: Present and moderate #(2-3 spasms) | 2 | 4 | 2 | 3
  Colonic Spasm WIthdrawal: Present and high # (4-5 spasms) | 2 | 0 | 0 | 1
  Colonic Spasm WIthdrawal: Present and very high (>5 spasms) | 0 | 0 | 0 | 0

8. Secondary Outcome: Patient's Willingness to Repeat Experience
Description: Patients' willingness for repeat colonoscopy, was assessed with the Patient Willingness to Repeat Experience (P.W.R.E.) questionnaire (1 question), asking patients to rate their willingness to repeat the procedure according to a 5-point Likert scale: Strongly Agree, Agree, Agree nor Disagree, Disagree, Strongly Disagree. The P.W.R.E was administered after the colonoscopy during subject recovery.
Time Frame: Post-colonoscopy- during subject recovery
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | GIC-1001 Low Dose | GIC-1001 Mid-dose | GIC-1001 , High Dose | GIC-1001 Matching Placebo
Number analyzed (Participants) | 56 | 52 | 53 | 101
Participants
  Strongly Agree | 23 | 26 | 15 | 42
  Agree | 16 | 17 | 18 | 32
  Agree nor Disagree | 8 | 2 | 5 | 11
  Disagree | 5 | 5 | 5 | 6
  Strongly Disagree | 4 | 2 | 8 | 8
  Missing | 0 | 0 | 2 | 2

9. Secondary Outcome: Subject Satisfaction and Acceptability of the Colonic Analgesia - Patient's Global Impression of Abdominal Pain
Description: Subject satisfaction and acceptability of the colonic analgesia modality offered by GIC-1001 was assessed with the Patient Global Impression of Abdominal Pain (P.G.I.A.P.) (1 question), asking patients to rate their pain during the procedure according to a 5-point Likert scale: Absent, Mild, Moderate, Severe, Intolerable. The P.G.I.A.P was administered after the colonoscopy during subject recovery.
Time Frame: Post-colonoscopy- during subject recovery
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | GIC-1001 Low Dose | GIC-1001 Mid-dose | GIC-1001 , High Dose | GIC-1001 Matching Placebo
Number analyzed (Participants) | 56 | 52 | 53 | 101
Participants
  Absent | 6 | 4 | 3 | 13
  Mild | 21 | 17 | 15 | 30
  Moderate | 17 | 21 | 22 | 29
  Severe | 12 | 7 | 8 | 21
  Intolerable | 0 | 3 | 3 | 6
  Missing | 0 | 0 | 2 | 2

ADVERSE EVENTS:
Time Frame: Assessed before drug treatment, on Day 2 of the 3-day dose regimen, before and after the colonoscopy (Day4), followed by 2 safety call after 48 hours post-colonoscopy and 7 days post-colonoscopy.
Description: Safety was assessed via performance of physical exams, vital signs, 12-lead ECG, laboratory safety tests (hematology, biochemistry and urinalysis) and the occurrence of adverse events.
Arm/Group | GIC-1001 Low Dose | GIC-1001 Mid-dose | GIC-1001 , High Dose | GIC-1001 Matching Placebo
All-Cause Mortality (participants affected / at risk) | 0/56 | 0/52 | 0/57 | 0/103
Serious Adverse Events (participants affected / at risk) | 0/56 | 0/52 | 0/57 | 0/103
Other Adverse Events (participants affected / at risk) | 46/56 | 41/52 | 48/57 | 85/103
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GIC-1001 Low Dose (N=56) | GIC-1001 Mid-dose (N=52) | GIC-1001 , High Dose (N=57) | GIC-1001 Matching Placebo (N=103)
Diverticulum (Gastrointestinal disorders) | 12 (68) | 10 (62) | 18 (65) | 22 (127)
Abdominal pain lower (Gastrointestinal disorders) | 3 (3) | 4 (5) | 5 (5) | 8 (9)
Haemorrhoids (Gastrointestinal disorders) | 14 (14) | 15 (15) | 15 (15) | 35 (35)
Nausea (Gastrointestinal disorders) | 6 (6) | 5 (5) | 5 (5) | 15 (17)
Large intestine polyp (Gastrointestinal disorders) | 10 (10) | 11 (11) | 9 (9) | 12 (12)
Polyp (General disorders) | 5 (5) | 2 (2) | 6 (6) | 9 (9)
Headache (Nervous system disorders) | 11 (11) | 9 (10) | 10 (11) | 20 (20)
Fatigue (General disorders) | 10 (10) | 5 (5) | 2 (2) | 10 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
this was stipulated in the contract